CLINICAL TRIAL: NCT06584656
Title: Understanding Cerebral Blood Flow Dynamics for Alzheimer's Disease Prevention Through Exercise: the flADex Study
Brief Title: Understanding Cerebral Blood Flow Dynamics for Alzheimer's Disease Prevention Through Exercise
Acronym: flADex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other); Instituto Mixto Universitario Deporte y Salud (iMUDS) (Unknown); Centro de InvestigaciÃ³n Mente, Cerebro y Comportamiento (Unknown)
Responsible Party: Principal Investigator, Irene Esteban-Cornejo, Ramon y Cajal Assistant Professor, PhD, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PID2022-137399OB-I0
Record Dates: First submitted 2024-08-06; First posted 2024-09-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy Aging; Cognitive Function 1, Social; Cerebrovascular Circulation; Blood Flow
Keywords: Alzheimer's Disease; Exercise; Cerebral Blood Flow; Biomarkers; Aging; Magnetic resonance imaging
MeSH Terms: conditions — Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise group (Experimental): -Aerobic group. 30 min at 60-70% of the Maximal Heart Rate, moderate intensity on cycle.
  Interventions: Behavioral: Aerobic exercise condition
- Resistance exercise group (Experimental): 30 min at 4-6 RPE (OMNI-Resistance Exercise Scale of Perceived Exertion), 3 sets of 8 exercise/set, 40 sec/exercise. Moderate intensity using elastic bands and body weight.
  Interventions: Behavioral: Resistance exercise condition
- Control (No Intervention): 30 min seated watching a neutral documentary without cognitive engagement

INTERVENTIONS:
Behavioral: Aerobic exercise condition — Aerobic session will last 30 min. The average intensity of the aerobic sessions will be 60-70% of the Maximal Heart Rate. Therefore, participant will perform a continuous moderate intensity aerobic bout of exercise on a cycle ergometer.
  Arms: Aerobic exercise group
Behavioral: Resistance exercise condition — Resistance exercise will last 30 min at 4-6 RPE (OMNI-Resistance Exercise Scale of Perceived Exertion from 0-10). The bout of resistance exercise will include a combination of upper and lower body exercises using elastic bands and the participants' body weight as the primary resistance. Eight different exercises will be performed per set, with 40 seconds per exercise, for a total of 3 sets. The exercises are based on basic movement patterns and include: glute bridge, front plank, standing face pull, incline push-up, squat, pallof press, walking lunge and seated shoulder press.
  Arms: Resistance exercise group

SUMMARY:
Dementia is one of the leading causes of disability worldwide. Underlying biological mechanisms are crucial in preclinical stages of Alzheimer's disease (AD). Alterations in cerebral blood flow (CBF) and their relationship with AD blood-based biomarkers may be fundamental at early stages of the pathology. Physical exercise is a trigger to modify these biological mechanisms. Therefore, flADex aims to examine the acute effects of different types of exercise (resistance vs. aerobic vs. control) on CBF, AD blood-based biomarkers, and its cognitive implications in older adults. The hypothesis is that acute resistance or aerobic exercise will fluctuate levels of blood-based biomarkers, and will exert acute CBF changes combined with cognitive implications.

DETAILED DESCRIPTION:
The aging population is at an increasing risk of developing Alzheimer's Disease (AD), which is characterized by cognitive decline and memory loss. Current pharmacological treatments have targeted amyloid-beta (Aβ) and tau protein, and have largely failed to halt or reverse the progression of AD. This has led to a growing interest on examining additional underlying mechanisms responsible for the initiation of AD pathology in this preclinical stage, such as cerebral blood flow (CBF) alterations or peripheral levels of AD blood-based biomarkers. Parallelly, exercise might act as a trigger for these potential underlying mechanisms of AD in older adults. Thus, this study seeks to explore the acute effects of different type of exercise on CBF, blood-based biomarkers, and its cognitive implications in older adults.

FlADex is a counterbalanced crossover trial that will include 20 adults aged 68 to 83 with non-pathological brain amyloid status (<12 centiloid) and APOE e4 noncarriers. Each participant will be included in all study conditions in a randomized order: (i) moderate aerobic exercise (between 60-70 of the Maximal Heart Rate (HRmax); (ii); resistance exercise (4-6 Moderate intensity of Rate of Perceived Exertion) and (iii) control resting condition. Each condition, lasting 30 minutes, will be performed once. CBF will be assessed by magnetic resonance imaging using pseudo-continuous arterial spin labeling at pre-condition and at 3 consecutive times post-condition (at 20', 27' and 34' min). Blood-based biomarkers (Aβ42, Aβ40, p-tau217, p-tau181, GFAP, NfL, BDNF, IGF-1) will be measured pre-condition and post-condition (at 0', 50', 70' min). Cognitive outcomes (Flanker Test and Picture Sequence Memory Test) and mood status (feeling scale and POMS questionnaire) will be measured pre and post condition.

FlADex trial will shed light on the acute effects of different types of exercises on CBF and AD blood-based biomarkers before beta-amyloid accumulation. We expect that aerobic and resistance exercise will have different effects on CBF dynamics and AD blood biomarker levels over time in older adults

ELIGIBILITY:
Inclusion Criteria:

* Older adults
* Aged 68-83 years
* Non-pathological cerebral beta-amyloid status (based on Centiloid cut-point <12 measured by PET-CT)
* APOEe4 negative status
* Willingness to participate in exercise interventions

Exclusion Criteria:

* Pathological diagnosis related to physical or mental condition
* No living in community settings during the study
* MRI incompatibility
* Ambulatory with pain or regular use of an assisted walking device
* Severe cardiovascular or respiratory conditions
* Participation in another clinical trial within the last 30 days

Ages: 68 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Change in Cerebral Blood Flow (CBF) | 30 minutes before the experimental condition; and 20 minutes, 27 minutes and 34 minutes minutes after the experimental condition
  Specific acquisition parameters for Pseudo continuous Arterial Spin Labeling (pCASL) sequence are used to determinate global and regional CBF in resting condition. Structural T1 sequence (only pre-condition) is used to coregisted the pCASL and delineate regions of interest for CBF. Time-of-flight angiography (TOF) (before pCASL pre-condition and before first pCASL post-condition) sequence is used to identify the carotid arteries. The unit of measurement of the CBF is expressed as milliliters per 100 grams of brain tissue per minute (mL/100 g/min).

SECONDARY OUTCOMES:
Change in Alzheimer disease blood-based biomarkers (Aβ42/40 ratio) | 5 minutes before the experimental condition; and 0 minutes, 50 minutes and 70 minutes after the experimental condition
  The following biomarkers will be assessed: Amyloid-beta 42 (Aβ42), Amyloid-beta 40 (Aβ40). Aβ42 and Aβ40 will be combined to report Aβ42/40 ratio. Unit of measurement: Aβ42/40 is a ratio (no units) and represents the relative concentration of Aβ42 to Aβ40.
Change in Alzheimer disease blood-based biomarkers (p-tau217, p-tau181, NfL and GFAP) | 5 minutes before the experimental condition; and 0 minutes, 50 minutes and 70 minutes after the experimental condition
  The following biomarkers will be assessed: phosphorylated tau protein at positions 217 and 181 (p-tau217, p-tau181), Glial Fibrillary Acidic Protein (GFAP) and Neurofilament Light Chain (NfL). Unit of measurement: p-tau217, p-tau181, NfL and GFAP are commonly measured in picograms per milliliter (pg/mL).
Change in growth factors (BDNF) | 5 minutes before the experimental condition; and 0 minutes, 50 minutes and 70 minutes after the experimental condition
  Brain-Derived Neurotrophic Factor (BDNF) will be measured. Unit of measurement: BDNF is commonly measured in picograms per milliliter (pg/mL).
Change in growth factors (IGF-1) | 5 minutes before the experimental condition; and 0 minutes, 50 minutes and 70 minutes after the experimental condition
  Insulin-Like Growth Factor 1 (IGF-1) will be measured. Unit of measurement: IGF-1 is commonly measured in nanograms per milliliter (ng/mL).
Change in episodic memory | 15 minutes before the experimental condition; and 60 minutes after the experimental condition
  Episodic memory will be assessed using the Picture Sequence Memory Test from the Cognitive NIH Toolbox. The Cognitive NIH Toolbox is a computer-based battery which is available in Spanish. The Picture Sequence Memory Test measures episodic memory by deriving the participant's score from the cumulative number of adjacent pairs of pictures remembered correctly over two learning trials. The variable used for the for the PSMT is the theta score: The number of adjacent pairs placed correctly for each of trials 1 and 2 is converted to a theta score. This is a representation of the given participant estimated ability in the task.
Change in inhibition/attention | 15 minutes before the experimental condition; and 60 minutes after the experimental condition
  The Flanker task measures inhibitory control and attention by using the inverse efficiency score of incongruent trials. The inverse efficiency score is calculated as reaction time/accuracy (RT/ACC).
Mood status | POMS will be measured 60 minutes before the experimental condition; and 70 minutes after the experimental condition
  Mood status will be evaluated using the validated scale Profile of Mood States (POMS). The POMS scale is a psychological assessment tool used to measure and evaluate a person's mood states. It consists of a questionnaire with a list of 15 adjectives or mood descriptors, where individuals rate how they have been feeling on a scale typically ranging from "Not at all" to "Extremely". We use an abbreviated version of the scale with 15 ítems. The ítems are divided into 5 dimensions: depression, vigour, anger, tension and fatigue. The final score is: ([depression]+[anger]+[tension]+[fatigue]) - [vigour].
Feeling scale | Feeling scale will be measured 1 minute before the experimental condition; and 1 minute after the experimental condition
  Emotional response will be evaluated using the feeling scale (FS). The FS is an 11-point scale ranging from -5 (very bad) to +5 (very good) used to measure an individual's emotional feeling in terms of pleasure or displeasure at a specific moment.

OTHER OUTCOMES:
Enjoyment | 5 minutes after the experimental condition
  Enjoyment of Physical activity will be assessed using the Physical activity Enjoyment scale (PACES): The PACES is an 18-item scale but we will use the reduced and validated version of 8 items, assessing in a range of 1 to 7 a series of sensations or moods with respect to its opposite, so that it is easier and more practical for participants.
Physical engagement (in aerobic condition and resistance condition) | During the experimental condition at minute 12, minute 20, and minute 30
  Perceived exertion of exercise (RPE) will be assessed using the OMNI-Resistance Exercise Scale (OMNI-RES) of perceived exertion from 0-10.
Repetitions in reserve (in resistance condition) | During the resistance condition after each exercise at minutes 5, 6, 7, 8, 9, 10, 11, 12 / 14, 15, 16, 17, 18, 19, 20, 21 / 23, 24, 25, 26, 27, 28, 29, 30
  The Repetitions in Reserve (RIR) will be assessed after each exercise in the resistance condition. RIR method is a self-regulation technique used in strength training to gauge exercise intensity. It involves estimating how many more repetitions you could perform before reaching failure after completing a set.
Cognitive engagement | During the experimental condition at minute 12, minute 20, and minute 30
  Cognitive engagement will be assessed by the Cognitive Load Measurement scale. The Cognitive Load Scale is a 9 ítem scale used to assess the mental effort or cognitive load experienced by individuals when engaging in a task, particularly in educational or learning contexts. It involves a self-reported measure where participants rate their perceived mental effort on a scale, ranging from 1 very low mental effort; to 9 very high mental effort.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Esteban-Cornejo, PhD, Principal Investigator — Department of Physical Education and Sports, Faculty of Sport Sciences, University of Granada, Spain.
Locations (2):
- Spain (2):
  - University of Granada, Granada, Andalusia
  - Mind, Brain, and Behaviour Research Centre (CIMCYC, Centro de Investigación Mente, Cerebro y Comportamiento), Granada

IPD SHARING:
Plan to Share IPD: Yes
The protocol, statistical analyses plan and data management plan will be sharing open access. Data files including IPD, and corresponding data dictionaries, will be shared under restricted access and upon reasonable request (contact Irene Esteban-Cornejo) due to privacy issue and GDPR regulations. In principle, all collected IPD will be available for sharing under the "as open as possible, as closed as necessary" principle. The shared data files will be pseudonymized, only include participants who provided informed consent for sharing, and sharing is only possible when the data is used for research purposes regarding exercise, and brain health. This is stated at the informed consent files that the participants signed when they agree to participate.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The IPD data will be available 12 months after the primary outcome paper published. The data will be available 15 years after data collection.
Access Criteria: The specific process of data access will be determined in a later stage, but in general the research team supports data sharing. Roughly, data will be available upon reasonable request to the PI (Irene Esteban-Cornejo). The data requests must contain the purpose and aim of the research, but also specification of the data requested, and data analysis before data sharing. Data will only be shared for research purposes on exercise and brain health. In addition, we will follow "as open as possible, as closed as necessary" principle, so depending on this principle we will decide whether the data could be shared. A data access committee will be installed to approve data requests.
URL: https://github.com/fladexprojectugr

REFERENCES:
- See also: Detailed information about the protocols, methodology , data analysis, and code used in this project will be upload to the GitHub repository: FLADEX Project GitHub Repository. — https://github.com/fladexprojectugr

DOCUMENTS (2):
  • Study Protocol (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT06584656/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT06584656/SAP_002.pdf